CLINICAL TRIAL: NCT04751344
Title: RANDOMIZED CONTROLLED TRIAL COMPARING LIPOSOMAL BUPIVACAINE VERSUS BUPIVACAINE HCL FOR POSTOPERATIVE MANAGEMENT OF FOREFOOT SURGERY
Brief Title: Liposomal Bupivacaine Versus Bupivacaine Plain for Operative Pain Management of Forefoot Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandra Black (Other)
Responsible Party: Sponsor-Investigator, Alexandra Black, DPM, Lenox Hill Hospital
Organization: Lenox Hill Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 101719
Record Dates: First submitted 2021-02-05; First posted 2021-02-12 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Liposomal Bupivacaine; Postoperative Pain; Forefoot Surgery; Opioid Use; Bunion
MeSH Terms: conditions — Pain, Postoperative; Bunion | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: Data will be encrypted using BRMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Liposomal Bupivacaine (Experimental): The liposomal bupivacaine study arm will receive 8cc (13.3 mg/mL) liposomal bupivacaine via intravenous route at the completion of the procedure.
  Interventions: Drug: Liposomal bupivacaine
- Bupivacaine HCl (Active Comparator): The Bupivacaine HCl study arm will receive 10cc (5mg/mL) of bupivacaine HCl via intravenous route at the completion of the procedure.
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Liposomal bupivacaine — Prior to procedure, surgeon will administer 15cc of Lidocaine 2% plain. After the procedure is finished, 8cc of liposomal bupivacaine (13.3mg/mL) will be injected around the surgical site.
  Other Names: Exparel
  Arms: Liposomal Bupivacaine
Drug: Bupivacaine HCl — Prior to procedure, surgeon will administer 15cc of Lidocaine 2% plain. After the procedure is finished, 10cc of bupivacaine HCl (5mg/mL) will be injected around the surgical site.
  Other Names: Marcaine
  Arms: Bupivacaine HCl

SUMMARY:
Prospective, randomized, controlled single-blinded trial comparing liposomal bupivacaine with bupivacaine HCl for postoperative management. Upon completion of the forefoot procedure in the operative room the subject will be entered into the randomization system which will specify whether to inject 10cc (5mg/mL) of bupivacaine HCl or 8cc (13.3 mg/mL) liposomal bupivacaine, both considered routine care procedure. Thereafter, postoperative pain will be assessed and measured using a Visual Analog Scale (VAS) scoring scale post-operatively at 2 hours, 24 hours, 48 hours and 72 hours. In addition, the amount of oral morphine equivalents (OME) required postoperatively and time to first use of OME will be measured. Our hypothesis is that patients who received liposomal bupivacaine will have less post-operative pain and require less OMEs.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, greater than 18 years of age
* ASA Class I or II
* Ability to take oral medication in order to assess the patient's opioid regimen postoperatively
* Forefoot surgery, including bunionectomy +/- digital surgery
* For females of reproductive potential: hCG levels will be determined during the pre-operative period. Females of childbearing age require a hCG level below 5mIU/mL in order to participate in the study. hCG levels above 25 mIU/mL is considered positive for pregnancy and, as a result, the patient will not be considered eligible for inclusion in the study

Exclusion Criteria:

* Chronic users of opioids, use for greater than 14 days in the last 3 months or nonopioid pain medications for more than 5 times per week
* Prescription for SSRIs, gabapentin, duloxetine within 3 days of surgery
* Systemic glucocorticoids within 1 month of study enrollment
* History of hepatitis
* History of peripheral vascular disease
* History of diabetes mellitus type 1 or 2
* Pregnancy or lactation
* Allergic to opioids
* Known allergic reactions to components of the bupivacaine injectable or other amide anesthetics; the allergen may involve preservative compounds such as methylparaben used in the preparation of amide-type agents are metabolized to PABA
* BMI > 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-16 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Effect of liposomal bupivacaine on postoperative pain control | The study will last 72 hours after the elective procedure.
  VAS scores, which measure the intensity of pain on a scale of 1 to 10, will be collected at 2, 24, 48 and 72 hours post-operatively in order to assess therapeutic effect of local anesthetic medication for postoperative pain control.

SECONDARY OUTCOMES:
Effect of liposomal bupivacaine on opioid use | The study will last 72 hours after the elective procedure.
  We will quantify opioid use post-operatively by collecting data on total opioid consumption and time to first use of the opioid post-operatively by the patient

CONTACTS AND LOCATIONS:
Overall Officials: Elliot Hershman, MD, Principal Investigator — Northwell Health
Locations (1):
- Manhattan Eyes Ears and Throat Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No